CLINICAL TRIAL: NCT03691064
Title: International, Non-interventional, Post-Authorization Long-Term Safety Study of Lutathera, in Patients With Unresectable or Metastatic, Well-Differentiated, Somatostatin Receptor Positive, Gastroenteropancreatic Neuroendocrine Tumours
Brief Title: Post-Authorization Long-Term Safety Study of LUTATHERA
Acronym: SALUS
Status: Active, not recruiting | Type: Observational
Sponsor: Advanced Accelerator Applications (Industry)
Responsible Party: Sponsor
Other Study IDs: A-LUT-T-E02-402; CAAA601A12402 (Other: Novartis); EUPAS25735 (Other: ENCePP)
Record Dates: First submitted 2018-09-22; First posted 2018-10-01 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-11

CONDITIONS: Neuroendocrine Tumors
Keywords: Gastroenteropancreatic neuroendocrine tumours
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — lutetium Lu 177 dotatate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LUTATHERA: Treated per labeled LUTATHERA dosing regimen.
  Interventions: Drug: LUTATHERA

INTERVENTIONS:
Drug: LUTATHERA — Labeled dosing regimen: 7.4 gigaBecquerel (GBq) (200 milliCurie [mCi]) every 8 weeks for a total of 4 doses.
  Other Names: Lu 177 dotatate

SUMMARY:
Study to assess the long-term safety of LUTATHERA for the labeled indication (SmPC/USPI).

DETAILED DESCRIPTION:
To assess the incidence and nature of potential long-term safety outcomes in patients with unresectable or metastatic, well-differentiated, somatostatin receptor positive gastroenteropancreatic neuroendocrine tumours. Retrospective and prospective data will be used.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (fulfilling the definition of "age of majority" per local regulations),
* with unresectable or metastatic, well-differentiated, somatostatin receptor positive GEP-NETs
* and who were treated with Lutathera (regardless of the quantity and number of doses administered and whatever the reasons for ending).

Exclusion Criteria:

* Hypersensitivity to Lutathera (active substance or any of the excipients),
* presence of established or suspected pregnancy or pregnancy not excluded,
* presence of kidney failure with creatinine clearance < 30 mL/min.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients treated with LUTATHERA for the labeled indication using the approved dosing regimen.
Sampling Method: Non-Probability Sample
Enrollment: 1014 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
secondary cancers: incidence of secondary cancers | up to 7 years follow-up
  incidence of secondary cancers

SECONDARY OUTCOMES:
safety profile: incidence of adverse events | up to 7 years follow-up
  incidence of adverse events
mortality | up to 7 years follow-up
  mortality (all cause)
LUTATHERA dose per administration | completion of treatment phase (approximately 2 years total)
  average dose per administration
LUTATHERA total dose | completion of treatment phase (approximately 2 years total)
  average total dose administered
LUTATHERA number of administrations | completion of treatment phase (approximately 2 years total)
  average number of LUTATHERA doses

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Advanced Accelerator Applications
Locations (17):
- United States (4):
  - Banner MD Anderson Cancer Center, Phoenix, Arizona
  - The Ohio State University Wexner Medical Center, Portland, Ohio
  - Oregon Health & Sciences University Hospital, Portland, Oregon
  - Virginia Mason in Seattle, Seattle, Washington
- France (3):
  - Novartis Investigative site, Clichy
  - Novartis Investigative site, Lyon
  - Novartis Investigative site, Villejuif
- Novartis Investigative site, Coimbra, Coimbra District, Portugal
- Spain (2):
  - Novartis Investigative site, Santiago de Compostela, La Corunya
  - Novartis Investigative site, Majadahonda, Madrid
- United Kingdom (7):
  - Novartis Investigative site, Birmingham
  - Novartis Investigative site, Cambridge
  - Novartis Investigative site, Glasgow
  - Novartis Investigative site, Liverpool
  - Novartis Investigative site, London
  - Novartis Investigative site, Manchester
  - Novartis Investigative site, Sheffield

IPD SHARING:
Plan to Share IPD: No